CLINICAL TRIAL: NCT03732924
Title: Zero to Five Automated Oscillometric Office Blood Pressure (AOBP) Measurement: the Impact of a 5 Minute Rest Time on AOBP Measurement
Brief Title: Zero to Five Automated Oscillometric Office Blood Pressure (AOBP) Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: KMH Cardiology and Diagnostic Centres (Other)
Responsible Party: Principal Investigator, Sheldon Tobe, Primary Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 181-2018
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Five minute rest (Experimental)
  Interventions: Diagnostic Test: Zero to Five Automated Oscillometric Office Blood Pressure (AOBP) Measurement
- Zero minute rest (Active Comparator)
  Interventions: Diagnostic Test: Zero to Five Automated Oscillometric Office Blood Pressure (AOBP) Measurement

INTERVENTIONS:
Diagnostic Test: Zero to Five Automated Oscillometric Office Blood Pressure (AOBP) Measurement — To compare the difference between the daytime ABPM and AOBP with zero or five minutes wait time.

SUMMARY:
The Hypertension Canada Clinical Practice Guidelines for blood pressure measurement using AOBP recommend against any wait time prior to commencing the measurement. The recent AHA guidelines however call for a 5-minute rest first. In uncontrolled hypertension, AOBP is typically higher than the daytime readings from ambulatory blood pressure monitoring (ABPM), but this is not the case for patients with controlled hypertension.

DETAILED DESCRIPTION:
Objective:

Does a 5 minute rest or no rest before measurement using AOBP provide the most accurate reading in patients with controlled and uncontrolled hypertension, and in patients with white coat hypertension compared to daytime ABPM?

Implications:

Through this study, we hope to:

(i) Advance the understanding of the role of AOBP in measuring blood pressure. (ii) Determine whether a 5-minute rest, or no rest at all is needed prior to AOBP measurement.

(iii) Assess the relationship of AOBP to daytime ABPM for patient with controlled and uncontrolled hypertension and in patients with white coat hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Referred for ABPM
* Written informed consent

Exclusion Criteria:

* Unable to perform AOBP or ABPM for some reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Difference in systolic and diastolic BP in patients randomized to zero or five minutes wait before the AOBP measurement. | 4 months - 1 yr
  difference in blood pressure

SECONDARY OUTCOMES:
Difference in systolic and diastolic BP between the AOBP and daytime ABPM in patients randomized to zero or five minutes wait before the AOBP measurement. | 4 months - 1yr
  difference in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon W Tobe, MD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobe SW, Dubrofsky L, Nasser DI, Rajasingham R, Myers MG. Randomized Controlled Trial Comparing Automated Office Blood Pressure Readings After Zero or Five Minutes of Rest. Hypertension. 2021 Aug;78(2):353-359. doi: 10.1161/HYPERTENSIONAHA.121.17319. Epub 2021 Jun 28. PMID 34176286